CLINICAL TRIAL: NCT05820035
Title: Focal Pulsed Field Ablation for Paroxysmal Supraventricular Tachycardia: A Prospective, Multicenter, Single-Arm Study in Mainland China
Brief Title: A Multicenter Study of Pulsed Field Ablation for Paroxysmal Supraventricular Tachycardia
Acronym: PSVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 775044
Record Dates: First submitted 2023-03-17; First posted 2023-04-19 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Paroxysmal Supraventricular Tachycardia; Atrioventricular Nodal Reentrant Tachycardia; Atrioventricular Reciprocating Tachycardia
Keywords: PFA; PSVT; AVNRT; AVRT
MeSH Terms: conditions — Tachycardia, Ventricular; Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental): Patients of PSVT treated with PFA catheter.
  Interventions: Device: Pulsed Field Ablation Device and CF-Sensing Pulsed Field Ablation Catheter

INTERVENTIONS:
Device: Pulsed Field Ablation Device and CF-Sensing Pulsed Field Ablation Catheter — All subjects will be ablated using the pulsed field ablation device and CF-sensing pulsed field ablation catheter in the management of their paroxysmal supraventricular tachycardia

SUMMARY:
The purpose of this study was to explore the safety and efficacy of pulsed field ablation（PFA) in the treatment of paroxysmal pupraventricular pachycardia（PSVT）with a contact force(CF)-sensing PFA Catheter

DETAILED DESCRIPTION:
The primary efficacy endpoints were to evaluate the acute and 6-month follow-up success rate after PFA without the use of antiarrhythmic drugs . The primary safety endpoints were to assess the incidences of serious adverse events (SAEs) at the end of the procedure , discharge and during the 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. age from 18 to 80 years,
2. episode of PSVT recorded by a 12-lead surface electrocardiogram (ECG), 24-hour Holter monitoring, or esophageal electrophysiologic study (EES) before hospitalization
3. reproducible clinical tachycardia confirmed by the electrophysiological study (EPS).

Exclusion Criteria:

1. Previous failure or recurrence of radiofrequency ablation
2. Left ventricular ejection fraction (LVEF) ≤ 40%
3. Combined with atrial flutter or atrial fibrillation
4. Combination of thromboembolic disease
5. Women who are breastfeeding, pregnant or planning to become pregnant during the study period
6. Carrying active implants in the body (e.g., pacemakers, ICDs, etc.)
7. Patients with second-degree (type II) or third-degree atrioventricular block
8. NYHA Class III-IV cardiac function [Appendix 1]
9. Patients with congenital heart disease (excluding atrial septal defect and patent foramen ovale)
10. Patients with definite acute cerebrovascular disease (including cerebral hemorrhage, stroke, transient ischemic attack) within the last 1 month
11. cardiovascular events within the last 3 months (including acute myocardial infarction, coronary intervention or heart bypass surgery, prosthetic valve replacement or repair, atrial or ventriculotomy)
12. Acute or severe systemic infection
13. Patients with severe liver and kidney diseases, malignant tumors and end-stage diseases
14. Patients with significant bleeding tendency, hypercoagulable state and serious hematologic disorders
15. Patients who have participated or are participating in other clinical trials within 3 months before enrollment
16. Patients who have other conditions that the investigator considers inappropriate for participation in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Primary efficacy and safety endpoints | at end of the procedure, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The primary efficacy endpoints were to evaluate the acute and 6-month follow-up success rate after PFA without the use of antiarrhythmic drugs. The primary safety endpoints were to assess the incidences of SAEs at the end of the procedure and during the 6-month follow-up period.

SECONDARY OUTCOMES:
Interim analysis | Refers to the postoperative phase after 6 months.
  To assess immediate ablation ablation success at 6 months postoperatively, by Holter in single center.

OTHER OUTCOMES:
Evaluation of Pulse Ablation equipment | immediately post ablation
  Whether the software can realize each set function, Whether the interface friendly and easy to operate, No abnormal software crash during the operation, et al.
Evaluation of Ablation voltage | immediately post ablation
  Record ablation voltage during ablation
Evaluation of Ablation sites | immediately post ablation
  Record ablation sites during ablation
Evaluation of Ablation x-ray time | immediately post ablation
  Record evaluation of Ablation x-ray time

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University (original name :Ningbo First Hospital), Ningbo, Zhejiang, China